CLINICAL TRIAL: NCT07075653
Title: Barriers to Adopting Vegetarian Diets Among Black and White Individuals With Chronic Medical Conditions
Brief Title: Barriers to Vegetarian Diets
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mihir Patel, Assistant Professor of Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00106683
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Chronic Disease
Keywords: vegetarian; vegetarian diet
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Midtown: This group includes participants recruited at the UMMC Midtown Campus.
  Interventions: Other: Survey using a questionnaire.
- UMMC: This group includes participants recruited at University of Maryland Medical Center.
  Interventions: Other: Survey using a questionnaire.
- UHC: This group includes participants recruited at the University of Maryland University Health Center.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — Participants fill out a brief survey in which they answer questions about vegetarian diets.

SUMMARY:
The goal of this observational study is to learn what affects a person's openness to adopting a vegetarian diet in urban community members with chronic disease.

The main questions it aims to answer are:

How open are individuals to adopting a vegetarian diet? What are the barriers to adopting a vegetarian diet?

Researchers will compare Black and White individuals to see if there are differences.

Participants will be asked to fill out a survey about their openness to going vegetarian as well as barriers to going vegetarian such as perceived stigma, tastiness, financial cost, convenience, familiarity, and healthfulness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-88 years old

Exclusion Criteria:

* Age <18 or >88 years old

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18-88 years old coming in for a clinic visit at one of 3 Baltimore hospitals/clinics.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Openness to going vegetarian | 5-10 minutes
  Openness is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Anticipated vegetarian stigma | 5-10 minutes
  Anticipated stigma is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Perceived tastiness of a vegetarian diet | 5-10 minutes
  Perceived tastiness is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Perceived financial cost of a vegetarian diet | 5-10 minutes
  Perceived financial cost is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Familiarity of a vegetarian diet | 5-10 minutes
  Familiarity is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Perceived convenience of a vegetarian diet | 5-10 minutes
  Perceived convenience is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).
Perceived healthfulness of a vegetarian diet | 5-10 minutes
  Perceived healthfulness is measured by the response to a set of statements on the survey where responses range from 1 (strongly disagree) to 7 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University Health Center, Baltimore, Maryland
  - University of Maryland Medical Center Midtown Campus, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No